CLINICAL TRIAL: NCT01733732
Title: Study to Evaluate the Efficacy of SYSTANE® BALANCE in Reducing Symptoms and Inflammatory Biomarker Expression of HLA-DR and Tear Film Cytokines in Dry Eye Subjects With Lipid Deficiency
Brief Title: SYSTANE® BALANCE Symptoms (OSDI) & Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00976
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2013-11

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye; Lipid deficiency; Inflammatory markers
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Balance (Experimental): SYSTANE® BALANCE Lubricant Eye Drops, 1 drop in each eye 4 times a day for 30 days
  Interventions: Other: SYSTANE® BALANCE Lubricant Eye Drops
- Systane Gel (Active Comparator): SYSTANE® Gel, 1 drop in each eye 4 times a day for 30 days
  Interventions: Other: SYSTANE® Gel

INTERVENTIONS:
Other: SYSTANE® BALANCE Lubricant Eye Drops
  Other Names: SYSTANE® BALANCE
  Arms: Systane Balance
Other: SYSTANE® Gel
  Arms: Systane Gel

SUMMARY:
The purpose of this study is to evaluate the ability of SYSTANE® BALANCE and SYSTANE® Gel to improve comfort in subjects with dry eyes.

ELIGIBILITY:
Inclusion Criteria:

* Read, sign, and date the Informed Consent Document;
* Must not have used any topical ocular drops for approximately 24 hours prior to Visit 1;
* Meet the protocol-specified dry eye criteria at Screening Visit (Visit 1);
* Intraocular pressure (IOP) less than or equal to 22 millimeters of mercury (mmHg) in both eyes;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery or serious trauma in either eye within the past 6 months;
* Current punctal occlusion of any type (e.g., collagen plugs, silicone plugs);
* History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye;
* Use of any concomitant topical ocular medications during the study period;
* Currently using Restasis but unwilling to discontinue its use 1 month prior to screening and for the entire study period;
* Use of systemic medications that may contribute to dry eye unless on a stable dosing regimen for a minimum of 30 days prior to Visit 1 and that remains stable throughout the study;
* Uncontrolled ocular conditions such as uveitis, glaucoma or any other ocular condition that may preclude the safe administration of either drop under investigation;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research; Penny A. Asbell, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the US.
Pre-assignment Details: A total of 54 subjects were screened and randomized. This reporting group includes all randomized subjects (54).
Groups:
- Systane Balance; Systane Gel: One drop in each eye 4 times a day for 30 days
Period: Overall Study
Arm/Group | Systane Balance | Systane Gel
Started | 27 | 27
Completed | 25 | 27
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Did not attend all study visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Balance | Systane Gel | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.5) | 63.8 (12.8) | 63.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Ocular Comfort Measured as Mean Change From Baseline in OSDI Score by Visit
Description: The Ocular Surface Disease Index (OSDI) is a 12-question validated questionnaire used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision. The OSDI scoring scale ranges from 0 to 100. The lower the score, the more symptomatic relief from dry eye symptoms a patient experiences. Baseline-adjusted scores were tabulated; a negative number change from baseline indicates a perceived improvement in ocular comfort.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: This analysis population includes all subjects who were randomized and attended at least one post-baseline study visit. Here, "n" is the number of subjects with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
units on a scale
  Change from baseline at Day 14, n=25, 27 | -7.85 (18.19) | -12.58 (19.05)
  Change from baseline at Day 30, n=27, 27 | -10.23 (21.72) | -16.74 (21.13)

2. Secondary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) by Visit
Description: BCVA (with spectacles or other visual corrective devices) was determined using an ETDRS or modified EDTRS chart and measured in logMAR (logarithm of the minimum angle of resolution). Baseline-adjusted logMAR values were tabulated; a negative number change from baseline indicates better visual acuity. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: This analysis population includes all subjects who were randomized and attended at least one post-baseline study visit. Here, "n" is the number of eyes with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
LogMAR
  Change from baseline at Day 14, n=50, 53 | -0.02 (0.06) | -0.01 (0.04)
  Change from baseline at Day 30, n=54, 51 | -0.02 (0.06) | -0.02 (0.06)

3. Secondary Outcome: Percentage of Eyes With Normal Slit-lamp Assessment
Description: An undilated slit lamp exam was performed to examine the regions of the eye: orbit/lids, conjunctiva, cornea, anterior chamber, iris and lens. Each region was graded normal or abnormal. The percentage of eyes with normal assessments by region is reported. Each eye was assessed individually. Both eyes were included in the tabulation.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: This analysis population includes all subjects who were randomized and attended at least one post-baseline study visit. The actual sample size used in calculating the outcome measure may be smaller due to missing responses and/or visit attendance.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Systane Balance, Day 0; Systane Balance, Day 14; Systane Balance, Day 30; Systane Gel, Day 0; Systane Gel, Day 14; Systane Gel, Day 30: One drop in each eye 4 times a day for 30 days
Arm/Group | Systane Balance, Day 0 | Systane Balance, Day 14 | Systane Balance, Day 30 | Systane Gel, Day 0 | Systane Gel, Day 14 | Systane Gel, Day 30
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Number analyzed (eyes) | 54 | 54 | 54 | 54 | 54 | 54
percentage of eyes
  Orbit / Lids | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Conjunctiva | 92.6 | 96.0 | 96.3 | 96.3 | 100.0 | 100.0
  Cornea | 92.6 | 92.0 | 92.6 | 92.6 | 92.6 | 92.6
  Anterior chamber | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Iris | 94.4 | 94.0 | 94.4 | 100.0 | 100.0 | 100.0
  Lens | 44.4 | 44.0 | 44.4 | 51.9 | 51.9 | 51.9

4. Secondary Outcome: Meibomian Gland Expression
Description: Meibomian gland expression (ie, pressing on the meibomian glands to excrete oil) was performed by the investigator during undilated slit lamp examination and graded on a 4-point scale where 0=normal, clear oil expressed and 3=congealed or no material expressed. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
units on a scale
  Baseline (Day 0), n=54, 54 | 1.4 (0.60) | 1.6 (0.77)
  Day 14, n=50, 54 | 1.2 (0.59) | 1.3 (0.59)
  Day 30, n=54, 54 | 1.2 (0.59) | 1.3 (0.68)

5. Secondary Outcome: Mean Change From Baseline in Non-invasive Keratographic Tear Break up Time (NIKBUT) by Visit
Description: NIKBUT (time required for dry spots to appear on the surface of the eye after blinking) was measured in seconds using the Oculus keratograph 5M. Baseline-adjusted scores were tabulated; a positive number change from baseline indicates improvement. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
seconds
  Change from baseline at Day 14, n=45, 54 | 0.587 (6.696) | -0.325 (4.557)
  Change from baseline at Day 30, n=49, 52 | -0.914 (5.697) | 1.261 (6.633)

6. Secondary Outcome: Mean Change From Baseline in Tear Meniscus Height (TMH) by Visit
Description: TMH (the distance between the line of reflection along the top of the tear prism to the edge of the eyelid) was measured in millimeters using the Oculus keratograph 5M. Baseline-adjusted scores were tabulated; a positive number change from baseline indicates improvement. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
millimeters
  Change from baseline at Day 14, n=50, 54 | 0.146 (0.165) | 0.089 (0.181)
  Change from baseline at Day 30, n=54, 52 | 0.140 (0.168) | 0.165 (0.242)

7. Secondary Outcome: Mean Change From Baseline in Ocular Surface Staining by Visit
Description: Ocular surface staining (damage to the ocular surface) was assessed using non-toxic ophthalmic dye during slit-lamp review. Corneal and conjunctival staining were graded as per the National Eye Institute (NEI) pictorial scale. The ocular staining score ranges from 0 to 3. The lower the score, the less signs of dry eye disease a patient exhibits. Baseline-adjusted scores were tabulated; a negative number change from baseline indicates an improvement. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Systane Balance, Change From Baseline at Day 14; Systane Balance, Change From Baseline at Day 30; Systane Gel, Change From Baseline at Day 14; Systane Gel, Change From Baseline at Day 30: One drop in each eye 4 times a day for 30 days
Arm/Group | Systane Balance, Change From Baseline at Day 14 | Systane Balance, Change From Baseline at Day 30 | Systane Gel, Change From Baseline at Day 14 | Systane Gel, Change From Baseline at Day 30
Number analyzed (Participants) | 25 | 27 | 27 | 27
Number analyzed (eyes) | 50 | 54 | 54 | 54
units on a scale
  Corneal staining | -1.0 (2.0) | -0.9 (2.3) | -1.3 (2.2) | -1.6 (2.4)
  Conjunctival staining | -0.7 (1.4) | -0.7 (1.4) | -0.9 (1.5) | -1.0 (1.4)

8. Secondary Outcome: Mean Change From Baseline in Tear Inflammatory Cytokine Expression at Day 30
Description: A tear sample was collected and cytokine (small proteins) levels were analyzed using a High Sensitive Human Cytokine MilliPlex kit and measured in picograms/milliliter (pg/mL). Baseline-adjusted scores were tabulated; a negative number change from baseline indicates improvement. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
pg/mL
  IFN-gamma, n=24, 25 | 2.680 (14.366) | 15.146 (65.229)
  IL-1beta, n=24, 25 | 0.192 (1.161) | 0.335 (2.515)
  IL-6, n=24, 25 | 0.902 (5.009) | 0.735 (16.364)
  TNF-alpha, n=24, 25 | -0.058 (1.713) | 0.693 (5.727)

9. Secondary Outcome: Mean Change From Baseline for % HLA-DR Inflammatory Biomarker Expression at Day 30
Description: Conjunctival samples were collected by Impression Cytology (IC) and analyzed in a lab. The number of cells expressing the inflammatory marker HLA-DR (as a percentage of total cells) was calculated. Baseline-adjusted scores were calculated as HLA-DR score at Day 30 minus HLA-DR score at baseline. A negative baseline-adjusted value indicates an improvement. Each eye was assessed individually. Both eyes were included in the mean.
Time Frame: Baseline (Day 0), Day 30
Population: This analysis population includes all subjects who were randomized and attended at least one post-baseline study visit.
Measure: Mean (Standard Deviation); unit: percentage of cells
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
percentage of cells | -0.751 (1.934) | -0.300 (0.844)

10. Secondary Outcome: Mean Change From Baseline mRNA for % HLA-DR and TNF-alpha Gene Expression at Day 30
Description: Conjunctival samples were collected by Impression Cytology (IC) and analyzed in a lab. Total RNA was isolated. The number of cells expressing the inflammatory marker (as a percentage of total cells) was calculated. Baseline-adjusted scores were calculated as score at Day 30 minus score at baseline. A negative baseline-adjusted value indicates an improvement. Each eye was assessed individually. Both eyes were included in the mean.
Time Frame: Baseline (Day 0), Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
percentage of cells
  HLA-DR, n=19, 25 | 0.079 (2.199) | 0.019 (1.027)
  TNF-alpha, n=20, 23 | -0.061 (0.313) | 0.009 (0.140)

11. Secondary Outcome: Mean Change From Baseline in Dry Eye Status as Measured by the Schirmer's Test by Visit
Description: Dry eye status was assessed using the Schirmer's test. The investigator placed a paper strip on the eye under the lower lid for a specified time period. The length of the strip wetted by the tears was measured in millimeters. Baseline-adjusted values were tabulated; a positive number change from baseline indicates an improvement. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
millimeters
  Change from baseline at Day 14, n=50, 54 | -0.3 (7.0) | 2.8 (7.9)
  Change from baseline at Day 30, n=54, 54 | 4.6 (8.5) | 2.6 (8.2)

12. Secondary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP) by Visit
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Baseline-adjusted values were tabulated. Each eye was assessed individually. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Systane Balance | Systane Gel
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 54 | 54
mmHg
  Change from baseline at Day 14, n=50, 54 | 0.0 (0.5) | 0.2 (0.9)
  Change from baseline at Day 30, n=54, 54 | 0.1 (1.4) | -0.1 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (7 months). This analysis group includes all subjects exposed to the test product.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Reports of AEs were obtained through volunteered and elicited comments from the subjects.
Arm/Group | Systane Balance | Systane Gel
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Systane Balance (N=27) | Systane Gel (N=27)
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.